CLINICAL TRIAL: NCT03708016
Title: Effect of Robot Gait Training With Brain Stimulation on Gait Function in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-05-015
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot gait training with brain stimulation (Experimental): Lokomat robot training and anodal transcranial direct current stimulation (tDCS) on the leg motor areas
  Interventions: Device: Robot gait training; Device: Brain stimulation
- Robot gait training without brain stimulation (Active Comparator): Lokomat robot training and sham tDCS on the leg motor areas
  Interventions: Device: Robot gait training

INTERVENTIONS:
Device: Robot gait training — Lokomat robot training was applied to stroke patients.
Device: Brain stimulation — tDCS brain stimulation on leg motor areas was applied to stroke patients.
  Arms: Robot gait training with brain stimulation

SUMMARY:
The purpose of this study was to investigate the effects of robot gait training with the noninvasive brain stimulation in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: more than 18 years
* More than 6 months post stroke
* Functional ambulation classification (FAC) (1~4)

Exclusion Criteria:

* Serious cardiac conditions (hospitalization for myocardial infarction or heart surgery within 3 months, history of congestive heart failure, documented serious and unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living)
* Difficult to understand experimental tasks because of extremely severe cognitive impairment
* History of disorders involving central nervous system
* History of psychiatric disease
* implanted objects that would contraindicate tDCS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Change in 10 meter walk test from baseline in gait speed | session 0 (initial visit); session 10 (at approximately 3 weeks); after 1 months from intervention termination (follow-up)
  Measure of self selected speeds by measuring the time it takes an individual to walk 10 meters. To perform the test, patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance at your normal pace when I say go."

SECONDARY OUTCOMES:
Change in Berg Balance Scale from baseline in balance | session 0 (initial visit); session 10 (at approximately 3 weeks); after 1 months from intervention termination (follow-up)
  Meserue of blance function
Change in Functional ambulatory category from baseline in gait function | session 0 (initial visit); session 10 (at approximately 3 weeks); after 1 months from intervention termination (follow-up)
  Measure of functional ambulatory category
Change in Timed Up and Go test from baseline in balance | session 0 (initial visit); session 10 (at approximately 3 weeks); after 1 months from intervention termination (follow-up)
  Measure of Timued Up and Go test in balance
Change on gait function (kinematic) | session 0 (initial visit); session 10 (at approximately 3 weeks); after 1 months from intervention termination (follow-up)
  All participants perform overground walking to assess the change of kinematic using a motion analysis.
Change on gait function (kinetic) | session 0 (initial visit); session 10 (at approximately 3 weeks); after 1 months from intervention termination (follow-up)
  All participants perform overground walking to assess the change of kinetic using a force plate
Change on gait function (muslce activation) | session 0 (initial visit); session 10 (at approximately 3 weeks); after 1 months from intervention termination (follow-up)
  All participants perform overground walking to assess the change of muscle activation using a surface EMG.
Changes in motor evoked potentia | session 0 (initial visit); session 10 (at approximately 3 weeks); after 1 months from intervention termination (follow-up)
  measure the motor threshold and amplitude of motor evoked potential in first dorsal interosseous muscle and TA muscle.
Changes in Brain activation of resting-state functional MRI | session 0 (initial visit); session 10 (at approximately 3 weeks); after 1 months from intervention termination (follow-up)
  Neuroplasticity measure

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided